CLINICAL TRIAL: NCT02011607
Title: Incidence of Adverse Airway Events in High Risk Patients Undergoing Upper GI Endoscopy Under Anesthesia
Acronym: SEDLine
Status: Terminated | Type: Observational
Why Stopped: Lack of support
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 812903
Record Dates: First submitted 2013-09-14; First posted 2013-12-13 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: SEDLine; Accoustic Respiratory Monitor RAD87; Adverse Events; Advanced Endoscopic Procedures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We propose to collect the data of vital signs and anesthesia medications administered in a subcategory of patients coming for anesthesia for upper GI endoscopy. This data will be analyzed to see any relation between the preoperative risk factors, procedure, type of anesthesia and the airway intervention. The adverse events that will be automatically recorded and later analyzed will be number of apnea episodes (described as no respiration for at least 30 seconds) duration of each apnea, number and duration of each desaturation event (oxygen saturation as measured by the pulse oximeter). A pulse oximeter saturation of less than 93 percent and lasting 30 seconds will be considered as a desaturation event. The airway interventions that will be recorded will be anything other than considered being routine. This includes LMA insertion, endotracheal intubation and the need to withdraw gastroscope to facilitate face mask ventilation. We also propose to monitor their awareness/depth of sedation/depth of anesthesia levels. This will be done using a monitor that analyses brain waves and gives an idea of sleep (anesthesia) depth. We can then see any correlation between any unwanted events and the sleep depth.

ELIGIBILITY:
Inclusion Criteria:

* All the patients considered as high risk (see above) or undergoing an advanced upper GI procedure (see above) will be included. This is the prospective analysis of the data that is collected and stored in the monitors. We will be using the massimo Pulse oximeter ,masimo acoustic respiratory monitor and Masimo SED line Brain function monitors that allows electronic storage and retrieval of information.
* Postprocedure analysis of the data will not influence the patient care.

Exclusion Criteria:

* Any patient who cannot give a valid consent will be excluded
* Children
* Pregnant women
* Fetuses and/or Neonates
* Prisoners

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patints undergoing advanced endoscopic procedures
Sampling Method: Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2013-01; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
incidence of adverse events | during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Basavana G Goudra, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of pennsylvania, Philadelphia, Pennsylvania, United States